CLINICAL TRIAL: NCT01622374
Title: a Randomized Controlled Clinical Trial on the Effects of "Music for the Mind" on Pre-operative Anxiety in Dentistry
Brief Title: Effects of "Music for the Mind" on Pre-operative Anxiety in Dentistry
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aminpasha Samadian, researcher in Azad University of Medical Sciences, Azad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Aminpasha_CT0001
Record Dates: First submitted 2012-06-14; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Dental Anxiety
Keywords: Music; dental anxiety; "music for the mind"; mozart; iranian traditional music
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Silence (Active Comparator): the subjects received 10 minutes of silence through headphone
  Interventions: Behavioral: Music
- Music for the mind (Experimental)
  Interventions: Behavioral: Music
- Mozart music (Experimental)
  Interventions: Behavioral: Music
- Iranian traditional music (Experimental)
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — Ten minutes of music or silence were applied prior to dental procedures
  Other Names: Music for the mind; Mozart Music; Iranian Music

SUMMARY:
To examine the pre-operative effect of music for the mind compared to some other styles of music in patients undergoing dental procedures.

DETAILED DESCRIPTION:
120 patients were sequentially assigned to four groups of 30 subjects. the music groups received Music for the mind, Iranian traditional music and Mozart music through headphone for ten minutes prior to dental procedures, and the control group received silence through headphone. anxiety score and pulse rate and blood pressure were measured before and after receiving music

ELIGIBILITY:
Inclusion Criteria:

* need for dental treatments

Exclusion Criteria:

* usage of anxiety drugs
* usage of psychoactive drugs
* emergency cases

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
STAI Inventory | 5 minutes
  The level of anxiety was measured by STAI Inventory index immediately after the intervention

SECONDARY OUTCOMES:
Heart rate | 30 seconds
  The index was measured before and after the intervention
Systolic blood pressure | 30 seconds
  The index was measured before and after the intervention
Diastolic blood pressure | 30 seconds
  The index was measured before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Aminpasha Samadian, DDS, Study Chair — Azad university of medical science